CLINICAL TRIAL: NCT04605029
Title: Frailty, Outcomes, Recovery and Care Steps of Critically Ill Patients - A Pilot Study
Brief Title: Frailty, Outcomes, Recovery and Care Steps of Critically Ill Patients
Acronym: FORECAST
Status: Completed | Type: Observational
Sponsor: Dr. John Muscedere (Other)
Collaborators: Canadian Frailty Network (Other)
Responsible Party: Sponsor-Investigator, Dr. John Muscedere, Critical Care Research Director, Queen's University
Organization: Queen's University (Other)
Other Study IDs: FORECAST
Record Dates: First submitted 2018-10-30; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Critical Illness
Keywords: Frailty
MeSH Terms: conditions — Critical Illness; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cytokine levels and measures of immunocompetence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically Ill patients: No Intervention

SUMMARY:
This pilot study will study the impact of critical illness and ICU processes of care on the trajectory and development of frailty. It is hypothesize that frailty in survivors of critical illness will be measurable at hospital discharge, will correlate with processes of care while in ICU and will better discriminate long term outcomes when compared to severity of illness or the degree of frailty present on ICU admission.

This pilot study will be conducted in a tertiary medical surgical ICU at Kingston General Hospital- Kingston, Ontario. It will inform the feasibility, timelines and sample size for the multi-center study and will allow for the refinement of study procedures and data collection methods. This study will be published separately as a stand-alone pilot.

DETAILED DESCRIPTION:
Single Center Observational pilot study to inform on the conduct of a multi-center observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 55 years
2. Admission to ICU for over 24 hours
3. Receipt of at least one therapeutic life support intervention that can only be delivered in the ICU such as mechanical ventilation (both invasive and non-invasive), vasoactive medications (vasopressors or inotropes) or acute renal replacement therapy.

Exclusion Criteria:

1. Lack of consent for study inclusion or lack of consent to be contacted for long term follow-up.
2. Expected to survive for less than 72 hours after ICU admission.
3. Inability to obtain baseline blood work less than 48 hours after ICU admission (i.e. study enrollment must occur within 48 hours of ICU admission allowing for the blood work to be done in the time allowed).
4. No family or caregivers available to collect collateral history.
5. Not able to speak English with lack of available medical translators.
6. Admission to ICU with acute structural neurological disease:

   1. Massive stroke requiring ICU care
   2. Spinal cord injury with neurological deficit

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who are admitted to an intensive care unit requiring therapeutic life support.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with a measure of frailty prior to hospital discharge. | 6 months
  Measure of the Frailty Index and Clinical Frailty Scale prior to discharge
Correlation of frailty severity at hospital discharge with long term outcomes (mortality, Quality of Life and Need for Institutionalization) | 6 months
  Clinical outcomes at 6 months will include mortality, Quality of Life (EQ5L) and need for Institutionalization
Impact of admission critical illness on the development and severity of frailty as measured by a Frailty Index or Clinical Frailty Scale | 28 days and at 6 months
  Correlation with the progression or presence of frailty as measured with the Frailty Index or Clinical Frailty Scale
Correlation of ICU processes of care (nutritional adequacy, mobilization and sedation) with frailty progression as measured by the Clinical Frailty Scale or Frailty Index | 28 days
  Correlation of processes of care in ICU (nutritional adequacy, mobilization and sedation) with frailty progression

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided